CLINICAL TRIAL: NCT02359409
Title: Use of Goggle Balloon to Improve Cecal Intubation During Colonoscopy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no subjects consented due to competing studies
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Douglas K. Rex, Director of Endoscopy, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IndianaU; NCT02539888 (obsolete NCT alias)
Record Dates: First submitted 2015-01-30; First posted 2015-02-10 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Redundant Colon

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- water immersion only (Active Comparator): Colonoscopy will be performed using the water immersion technique.
  Interventions: Other: water immersion only
- water immersion with goggle balloon (Experimental): Colonoscopy will be performed using a goggle balloon at the tip of the scope with water immersion technique
  Interventions: Device: goggle balloon

INTERVENTIONS:
Device: goggle balloon — Colonoscopy will be performed using the water immersion technique.
  Arms: water immersion with goggle balloon
Other: water immersion only — Colonoscopy will be performed using a goggle balloon at the tip of the scope with water immersion technique.
  Arms: water immersion only

SUMMARY:
This study aims to look if use of goggle balloon can help to complete colonoscopy in patients with very redundant colons.

DETAILED DESCRIPTION:
About 5% of colonoscopies are technically difficult because the colon is elongated or redundant. There is an increased risk of the colonoscope not reaching the cecum in these cases. One solution to this is to try to keep the colon shorter by not insufflating it with gas. In order to achieve that, in these cases the investigators typically fill the colon with water, which does not distend the colon as much. Another technique, which can improve visualization, is to use a device called the goggle balloon. This is a small balloon filled with a few mL of water which fits over the end of the colonoscope and pushes the colonic mucosa away from the end of the scope so that the luminal direction can be visualized with minimal insufflation. In patients with normal colons, the goggle balloon can be used to insert the colonoscope to the cecum with virtually no air or water filling. We aim to study if the goggle balloon can be used to help complete the colonoscopy in patients with redundant colons.

ELIGIBILITY:
Inclusion Criteria:

Referral for incomplete colonoscopy

Exclusion Criteria:

Known stricture or narrowing of the colon, prior colon resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2017-03-28 (Actual); Study Completion 2017-03-28 (Actual)

PRIMARY OUTCOMES:
number of subjects with complete colonoscopy in each arm | 2 years

SECONDARY OUTCOMES:
Time to cecal intubation in each arm | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Douglas K Rex, MD, Principal Investigator — IU Medical Center
Locations (1):
- Indiana University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No